CLINICAL TRIAL: NCT01762670
Title: An Open-Label, Randomized Study to Determine the Safety and Efficacy of GoldenCareTM for the Treatment of Bacterial Vaginosis
Brief Title: GoldenCareTM for the Treatment of Bacterial Vaginosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company decided to stop study for reasons other than safety
Sponsor: CDA Research Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDA 1106
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2013-07

CONDITIONS: Bacterial Vaginosis
Keywords: Bacterial Vaginosis; BV
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metronidazole (Active Comparator): Oral administration of metronidazole, 500 mg twice daily for 7 consecutive days
  Interventions: Drug: Metronidazole
- GoldenCare (Experimental): GoldenCare administered intravaginally for at least 6 hours at night for 7 consecutive nights.
  Interventions: Drug: GoldenCare

INTERVENTIONS:
Drug: GoldenCare — Copper intravaginal device to treat bacterial vaginosis.
  Other Names: Copper intravaginal device
  Arms: GoldenCare
Drug: Metronidazole — 500 mg twice daily for 7 days
  Other Names: Comparator
  Arms: Metronidazole

SUMMARY:
GoldenCare is a copper intravaginal device that may be useful for the treatment of symptomatic bacterial Vaginosis (BV). Standard treatment for BV is metronidazole. Although the reported cure rate is as high as 90%, the recurrence rate is 58% after 12 months. The study hypothesis is that GoldenCare will cure BV. This is a proof of concept study to collect preliminary evidence of the safety and efficacy of GoldenCare.

DETAILED DESCRIPTION:
GoldenCare is a copper intravaginal device that may be useful for the treatment of symptomatic bacterial Vaginosis(BV). Standard treatment for BV is metronidazole. Although the reported cure rate is as high as 90%, the recurrence rate is 58% after 12 months. The study hypothesis is that GoldenCare will cure BV. This is a proof of concept study to collect preliminary evidence of the safety and efficacy of GoldenCare.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Female aged 18 years or older
* Subject has clinical bacterial Vaginosis with 4 of 4 positive Amsel's criteria
* Negative pregnancy test
* For 7 day treatment period, subject agrees to refrain from using douches and intravaginal products (i.e. feminine deodorant sprays, spermicides, Nonoxynol-9 products, tampons, and condoms). Subject also agrees to refrain from taking oral or intravaginal antibiotics (unless enrolled in comparator arm),or antifungal agents during the entire study period.

Exclusion Criteria:

* Subject has another infectious or noninfectious cause of vulvovaginitis such asymptomatic candidiasis, Trichomonas vaginalis, Chlamydia trachomatis, Neisseria gonorrhoeae, Herpes simplex, human papilloma virus, atrophic vaginitis, lichen sclerosus, or genital warts.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of treating BV with GoldenCare for 7 days | 21 days
  Successful clinical cure of BV is defined as all 4 Amsel's criteria negative at Visit 4 and a Nugent score of 0-3 at Visit 4. Success will be determined at 21 to 30 days after first treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Chatwani, MD, Principal Investigator — Temple University Hospital Department of OB/GYN
Locations (2):
- United States (2):
  - Harper University Hospital Department of Infectious Diseases, Detroit, Michigan
  - Temple University Hospital Department of OB/GYN, Philadelphia, Pennsylvania